CLINICAL TRIAL: NCT03974347
Title: New Methods for Early Detection of Acute Kidney Injury After Heart Surgery
Status: Withdrawn | Type: Observational
Why Stopped: Logistical problmens, collisions with other studies
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Max Bell, Associate Professor, Karolinska Institutet
Other Study IDs: 2019-02319
Record Dates: First submitted 2019-06-02; First posted 2019-06-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Acute Kidney Injury
Keywords: cardiac surgery; renal resistive index; creatinine clearance
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine samples will be obtained. The following biomarkers will be measured NGAL, TIMP-2, IGFBP7, KIM-1, IL-18, L-FABP, cystatin C och angiotensinogen. Renal function markers Creatinine and urea will also be measured.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury, no acute kidney injury: Acute kidney injury after cardiac surgery will be defined by KDIGO criteria, Creatinine rise from baseline and or urine production.
- No Acute Kidney Injury: No Acute kidney Injury after Cardiac surgery, according to KDIGO AKI definition

SUMMARY:
The investigators intend to study 2 new methods for the early detection of Acute Kidney Injury (AKI) after cardiac surgery and compare and combine the predictive abilities of these methods with established renal injury markers and epidemiological models to detect (AKI).

DETAILED DESCRIPTION:
Acute Kidney Injury is common after Cardiac surgery and occurs in up to 20% of patients (Ref Rydén).

This study will evaluate two new methods for the early detection of acute kidney injury in 200 patients undergoing elective cardiac surgery at the Karolinska Hospital.

These methods are:

1. Ultrasound based measurement of the kidneys blood flow profile measured using renal resistive index (RRI). This will be measured prior and within 4 hours post surgery. Ref Herzberg, Le Dorze.
2. Urine creatinine clearance will be measured in the first four hours after cardiac surgery.

The investigators will also measure known renal injury markers in blood and urine samples post operatively. These include Neutrophil gelatinise-associated lipocalin (NGAL), tissue inhibitor of metalloproteinases (TIMP-2), Insulin-like growth factor-binding protein 7 (IGFBP7), Kidney Injury Molecule 1 (KIM-1), Nephroclear, Interleukin 18 (IL-18), Fatty acid-binding protein (L-FABP), Fibulin-1, cystatin C och albumin.

The new methods of AKI detection will be used to build a statistical model to predict AKI after cardiac surgery. We will determine whether the addition of renal injury markers and epidemiological factors known to be associated with the development of AKI (variables such as age, known chronic renal dysfunction or heart failure) can improve precision in diagnosis.

AKI will be defined by the Kidney Disease improving Global outcomes (KDIGO) criteria (Ref KDIGO KDIGO Clinical Practice Guideline for Acute Kidney Injury, Khwaja A).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Undergoing elective cardiac surgery (Coronary artery bypass grafting, valve surgery, aortic surgery or a combination).
* Able to understand and give written consent to partake in the study

Exclusion Criteria:

* Unable to give consent
* Previously received a renal transplant
* Renal failure requiring dialysis prior to surgery
* Persistent atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective cardiac surgery patients undergoing surgery at Karolinska University Hospital, Sweden. Patients with high risk for AKI as identified by the Clevland Clinic acute renal failure score will be identified.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 48 hours
  Acute Kidney Injury defined by KDiGO criteria

SECONDARY OUTCOMES:
30 day Mortality | 30 days
  Death occurring up to 30 days after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Max Bell, MD, PHD, Principal Investigator — Karolinska Institutet; Daniel Hertberg, MD, PHD, Study Director — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: Undecided
If the study data set is released it will be anonymized so that no personal data is retained and no individual can be identified from the data by those outside of the study.

REFERENCES:
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Le Dorze M, Bougle A, Deruddre S, Duranteau J. Renal Doppler ultrasound: a new tool to assess renal perfusion in critical illness. Shock. 2012 Apr;37(4):360-5. doi: 10.1097/SHK.0b013e3182467156. PMID 22258233
- [Background] Ryden L, Ahnve S, Bell M, Hammar N, Ivert T, Sartipy U, Holzmann MJ. Acute kidney injury after coronary artery bypass grafting and long-term risk of myocardial infarction and death. Int J Cardiol. 2014 Mar 1;172(1):190-5. doi: 10.1016/j.ijcard.2014.01.013. Epub 2014 Jan 22. PMID 24502882
- [Background] Hertzberg D, Ceder SL, Sartipy U, Lund K, Holzmann MJ. Preoperative Renal Resistive Index Predicts Risk of Acute Kidney Injury in Patients Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):847-852. doi: 10.1053/j.jvca.2016.10.006. Epub 2016 Oct 11. PMID 28017677
- [Background] Ryden LC, Sartipy U, Holzmann MJ. Acute Kidney Injury After Surgical AVR and Long-Term Risk of Death and End-Stage Renal Disease. J Am Coll Cardiol. 2015 Nov 17;66(20):2263-2264. doi: 10.1016/j.jacc.2015.08.883. No abstract available. PMID 26553408